CLINICAL TRIAL: NCT00790517
Title: Reducing Weight and Diabetes Risk in an Underserved Population
Brief Title: Reducing Weight and Diabetes Risk in an Underserved Population (STRIDE)
Acronym: STRIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); LifeWorks Northwest (Unknown); Cascadia Behavioral Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R18DK076775 (NIH); R18DK076775 (NIH); NCT00866372 (obsolete NCT alias)
Record Dates: First submitted 2008-09-12; First posted 2008-11-13 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Weight Loss; Diabetes Mellitus, Type 2; Psychotic Disorders
Keywords: Weight loss; Diabetes prevention; Serious mental illness; Antipsychotic medications; Lifestyle intervention; Antipsychotic Agents
MeSH Terms: conditions — Weight Loss; Diabetes Mellitus, Type 2; Psychotic Disorders | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Premier Lifestyle Intervention with Dash Diet, adapted for populations with mental illnesses
  Interventions: Behavioral: Premier Lifestyle Intervention with DASH Diet
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Premier Lifestyle Intervention with DASH Diet — Comprehensive group lifestyle intervention focused on caloric restriction and increased moderate exercise using the DASH Diet. 6 months intensive intervention (weekly, group meetings) followed by 6 months of a less-intensive maintenance intervention (monthly group meetings with monthly telephone/e-mail consult)
  Other Names: DASH Diet
  Arms: 1

SUMMARY:
The purpose of this study is to examine the effectiveness of a lifestyle intervention designed to reduce weight and diabetes risk in a population of individuals with mental illness who are also taking antipsychotic medications. We will examine the effectiveness of the intervention in

1. reducing weight and Body Mass Index;
2. reducing fasting insulin levels and increasing insulin sensitivity; and
3. reducing total cholesterol and LDL cholesterol.

DETAILED DESCRIPTION:
Overweight and obesity are among the leading causes of preventable deaths in the US, primarily through their effects on Type II diabetes mellitus and other cardiovascular disease risk factors. Individuals with serious mental illness represent a large underserved population at greatly increased risk of obesity, diabetes, metabolic syndrome, and subsequent early mortality. These risks are amplified by the antipsychotic agents that are often prescribed to treat these mental conditions.

Although strong evidence indicates that lifestyle interventions are effective at reducing weight and other diabetes risk factors in general populations, and pilot and feasibility studies suggest that such interventions will be effective with individuals who have mental illnesses, no large-scale translational trials have examined such interventions in this population.

STRIDE is a randomized controlled trial to examine the effectiveness, in a mentally ill population, of a lifestyle intervention previously shown to be effective for reducing weight and diabetes risk factors. We target a group of individuals taking antipsychotic agents (n = 280) who receive treatment in one of two clinical settings-a publicly funded behavioral health care clinic and a non-profit private health plan. Counselors from each clinical setting will be trained in the intervention and paired with study staff to deliver it, increasing generalizability, and improving the probability of future adoption. The intervention promotes moderate calorie reduction, dietary changes, and increased energy expenditure, and is based on current clinical practice guidelines for treating obesity and cardiovascular disease.

Specific aims test the hypotheses that the intervention is more effective than usual care in: 1) reducing weight and Body Mass Index; 2) reducing fasting insulin levels and increasing insulin sensitivity; and 3) reducing total cholesterol and LDL cholesterol. A fourth aim explores effects of motivation, social support, and outcomes expectancies on primary outcomes, and moderators of intervention effectiveness (ethnicity, gender, mental illness diagnostic group, medication type, metabolic syndrome) on outcomes.

Implementation and process evaluations will assess the fidelity of intervention delivery, evaluate its acceptability; identify components participants find most and least helpful; identify barriers to, and facilitators of, lifestyle changes; and evaluate the effects of the intervention on body image, psychiatric symptoms, adherence to antipsychotic medications, quality of life, health-related self-efficacy, health, functional status, and social support. Cost-effectiveness analyses will evaluate incremental costs of producing change in each primary outcome (weight, BMI, fasting insulin levels, insulin sensitivity, and cholesterol).

ELIGIBILITY:
Inclusion Criteria:

1. age 18 and over
2. stable on antipsychotic agents >1 month
3. BMI in the range of 25-44.9 kg/m2
4. approved by primary care provider or psychiatrist for participation (based on mental and physical health status)
5. able and willing to provide informed consent
6. access to telephone or e-mail (for maintenance phase)

Exclusion Criteria:

1. children under age 18
2. diagnosis of dementia
3. psychiatrist or primary care provider indication of any medical or psychiatric contraindications for participating in a weight reduction/exercise program
4. cardiovascular event within the past 6 months (if more remote history, eligible with primary care provider or psychiatrist approval)
5. history of bariatric surgery
6. cancer diagnosis or cancer treatment in the prior 2 years (except for non-melanoma skin cancer)
7. currently pregnant or breastfeeding, or plan a pregnancy prior to the end of study participation
8. mental health hospitalization in the 30 days prior to enrollment
9. planning on moving out of the area before the 24-month follow-up assessment
10. currently enrolled in a weight-reduction program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 6, 12, 24 months
Weight | 6, 12, 24 months
Insulin sensitivity | 6, 12, 24 months
Fasting insulin levels | 6, 12, 24 months
Cholesterol levels | 6, 12, 24 months

SECONDARY OUTCOMES:
Body Image | 6, 12, 24 months
Antipsychotic Medication Adherence | 6, 12, 24 months
Psychiatric Symptoms | 6, 12, 24 months
Health-related self-efficacy | 6, 12, 24 months
Social support for diet/weight loss | 6, 12, 24 months
Quality of life | 6, 12, 24 months
Health/functional status | 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Carla A Green, PhD, MPH, Principal Investigator — Center for Health Research, Kaiser Permanente Northwest
Locations (3):
- United States (3):
  - Cascadia Behavioral Healthcare, Portland, Oregon
  - Center for Health Research, Kaiser Permanente Northwest, Portland, Oregon
  - LifeWorks Northwest, Portland, Oregon

REFERENCES:
- [Derived] Yarborough BJ, Leo MC, Yarborough MT, Stumbo S, Janoff SL, Perrin NA, Green CA. Improvement in Body Image, Perceived Health, and Health-Related Self-Efficacy Among People With Serious Mental Illness: The STRIDE Study. Psychiatr Serv. 2016 Mar;67(3):296-301. doi: 10.1176/appi.ps.201400535. Epub 2015 Nov 2. PMID 26522674
- [Derived] Green CA, Yarborough BJ, Leo MC, Yarborough MT, Stumbo SP, Janoff SL, Perrin NA, Nichols GA, Stevens VJ. The STRIDE weight loss and lifestyle intervention for individuals taking antipsychotic medications: a randomized trial. Am J Psychiatry. 2015 Jan;172(1):71-81. doi: 10.1176/appi.ajp.2014.14020173. Epub 2014 Oct 31. PMID 25219423
- [Derived] Yarborough BJ, Leo MC, Stumbo S, Perrin NA, Green CA. STRIDE: a randomized trial of a lifestyle intervention to promote weight loss among individuals taking antipsychotic medications. BMC Psychiatry. 2013 Sep 28;13:238. doi: 10.1186/1471-244X-13-238. PMID 24074269